CLINICAL TRIAL: NCT03338309
Title: Multicenter Registry for Instantaneous Wave-Free Ratio (iFR)-Guided Percutaneous Coronary Intervention in Routine Clinical Practice
Brief Title: INsTantenous wavE-Free Ratio-guided PCI Versus Fractional Flow REserve-Guided PCI in rouTine Clinical Practice, Prospective, Multicenter Registry
Acronym: INTERPRET
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: NCT104658359911
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Stable Angina; Non ST Segment Elevation Myocardial Infarction; ST-segment Elevation Myocardial Infarction; Silent Myocardial Ischemia; Unstable Angina
Keywords: Fractional flow reserve; Instantaneous wave-free ratio; Ischemic heart disease
MeSH Terms: conditions — Angina, Stable; ST Elevation Myocardial Infarction; Angina, Unstable; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iFR-guied strategy group: 1,200 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, non ST-segment elevation MI, or ST-segment elevation MI with non-culprit stenosis who underwent iFR measurement and enrolled at 5 centers in Republic of Korea.
  Interventions: Other: Instantaneous wave-free ratio measurement

INTERVENTIONS:
Other: Instantaneous wave-free ratio measurement — Instantaneous wave-free ratio measurement in order to evaluate functional significance of epicardial stenosis

SUMMARY:
The current study sought to evaluate the clinical relevance of iFR-guided strategy in real world clinical practice using unrestricted study population from stable angina to acute coronary syndrome including acute ST-segment elevation myocardial infarction. Previous abundant historical data of FFR-guided strategy will be also included as historical control to validate the iFR-guided strategy.

DETAILED DESCRIPTION:
In this study, the investigators will validate the clinical relevance of instantaneous wave free ratio (iFR)-guided strategy in real world clinical practice in Korea. The 1,200 patients who underwent iFR measurement will be prospectively enrolled at 5 centers in Republic of Korea. In patients who were indicated revascularization after iFR measurement (iFR<0.90), iFR pullback system (iFR Scout) and post-revascularization iFR measurement will be routinely performed. The primary hypothesis will be tested for non-inferiority of iFR-guided strategy, compared with FFR-guided strategy in terms of 2-year clinical outcomes. For the clinical outcome data following FFR-guided strategy will be used from the pooled data of the DEFER-DES trial, the 3V FFR FRIENDS registry (NCT01621438), and Korean 4-center FFR registry. Using those data, 1200 patients will be selected from the pooled data. In addition, routine application of iFR Scout and post-revascularization iFR measurement will enable us to validate the clinical relevance of iFR-based prediction of acute procedural results and to compare FFR-pullback methods.

Primary Hypothesis: The iFR-guided strategy will be non-inferior regarding patient-oriented composite outcomes (a composite of any death, any MI, any revascularization) at 2-year, compared with FFR-guided strategy.

Primary Outcome:

1] Patient-oriented composite outcome (POCO), defined as a composite of any death, any myocardial infarction (MI) or any revascularization at 2-year after index procedure according to the ARC consensus [2] Difference between Predicted post-PCI iFR value from iFR Scout and Actual post-PCI iFR measurement

Sample Size 1,200 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, non ST-segment elevation MI, or ST-segment elevation MI with non-culprit stenosis enrolled at 5 centers in Republic of Korea.

1. Inclusion Criteria

   ① Subject must be ≥18 years

   ② Patients suspected with ischemic heart disease

   ③ Patients with coronary artery stenosis with intermediate degree of stenosis (40-70% stenosis by visual estimation) in major epicardial coronary artery amenable to stent implantation or vessel size≥2.5 mm without definitive previous evidence of myocardial ischemia.

   ④ Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and he/she or his/her legally authorized representative provides
2. Exclusion criteria

   * Cardiogenic shock (systolic blood pressure < 90mmHg or requiring inotropics to maintain blood pressure > 90mmHg) ② Patients with a known hypersensitivity or contraindication to any of the following medications: statin, ezetimibe, heparin, aspirin, clopidogrel, prasugrel, ticagrelor

     * Non-cardiac co-morbid conditions are present with life expectancy <2 year (per site investigator's medical judgment).

       * History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia) ⑤ Patients with active pathologic bleeding ⑥ Gastrointestinal or genitourinary major bleeding within the prior 3 months. ⑦ Target lesion located in coronary arterial bypass graft

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years

  * Patients suspected with ischemic heart disease ③ Patients with coronary artery stenosis with intermediate degree of stenosis (40-70% stenosis by visual estimation) in major epicardial coronary artery amenable to stent implantation or vessel size≥2.5 mm without definitive previous evidence of myocardial ischemia.

    * Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and he/she or his/her legally authorized representative provides

Exclusion Criteria:

* Cardiogenic shock (systolic blood pressure < 90mmHg or requiring inotropics to maintain blood pressure > 90mmHg)

  * Patients with a known hypersensitivity or contraindication to any of the following medications: statin, ezetimibe, heparin, aspirin, clopidogrel, prasugrel, ticagrelor ③ Non-cardiac co-morbid conditions are present with life expectancy <2 year (per site investigator's medical judgment).

    * History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia)

      * Patients with active pathologic bleeding ⑥ Gastrointestinal or genitourinary major bleeding within the prior 3 months. ⑦ Target lesion located in coronary arterial bypass graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,200 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, non ST-segment elevation MI, or ST-segment elevation MI with non-culprit stenosis who underwent iFR measurement and enrolled at 5 centers in Republic of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcome (POCO) | at 2-year after index procedure
  a composite of any death, any myocardial infarction (MI) or any revascularization according to the ARC consensus

SECONDARY OUTCOMES:
Difference between Predicted post-PCI iFR value from iFR Scout and Actual post-PCI iFR measurement | Immediate after post revascularization
  Difference between Predicted post-PCI iFR value from iFR Scout and Actual post-PCI iFR measurement

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — Seoul National University Hospital; Bon-Kwon Koo, MD, PhD, Study Director — Seoul National University Hospital; Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request after thorough discussion in steering committee